CLINICAL TRIAL: NCT03988491
Title: Predicting Morbidity, Mortality, Short and Long-term Survival of End-stage Kidney Disease Patients on Hemodialysis in Central Tanzania; a Two-center Prospective Patient-registry Observational Study.
Brief Title: Morbidity, Mortality, Short and Long-term Survival of Hemodialysis End-stage Kidney Disease Patients in Central Tanzania
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benjamin Mkapa Hospital (Other)
Responsible Party: Principal Investigator, Joel Dominic Swai, MD, Resident Physician-Internal Medicine Department, Benjamin Mkapa Hospital
Other Study IDs: BMH/J:89/30/VOL.X/2020
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: End-Stage Renal Disease
Keywords: Kidney Failure, Chronic; Mortality; Survival; Observational Study; Incidence; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End stage renal disease on maintanance hemodialysis: End-stage renal disease due to any etiology on maintenance hemodialysis and consented to participate in the study.

SUMMARY:
Background: In the last 2 decades, Tanzania made great improvements in the renal replacement therapy infrastructure and services. However, renal replacement therapy remains a challenge in the developing world in terms of inadequate renal registries, and limited published literature.

Objectives: This study will identify predictors of mortality, identify common causes of infection and hospitalization, their incidences, prevalence, and time-to-event analysis and analyze short and long-term survival of end-stage renal disease (ESRD) patients on hemodialysis in two hemodialysis centers in Dodoma, Tanzania. Furthermore, this study will establish a registry to be called Tanzania Registry for Chronic Renal Failure (TRCRF).

Methodology: This will be a prospective-observational study (Patient registry). It will be conducted in Tanzania, a developing world country involving two hemodialysis centers, namely Benjamin Mkapa Hospital and UDOM Health center, both affiliated with the University of Dodoma. Data will be collected by accessing patients' records receiving hemodialysis due to ESRD in the two centers from September 2019 to September 2024. Patients' demographics, medical history, investigation findings, and hemodialysis adequacy will be extracted as independent outcomes. In contrast, the outcome (i.e., Death) during the follow-up will be extracted as a primary dependent outcome. Binary logistic regression will be applied to come up with statistically significant predictors of deaths. Other outcomes will be incidences, prevalence, and time-to-event analysis of common causes of infection and re-hospitalization. Kaplan-Meier survival curves will be constructed from statistically significant predictors of deaths, and patients' survival at 1, 3, and 5 years will be illustrated.

DETAILED DESCRIPTION:
1. Background

   1.1 End-stage renal disease:

   End-stage renal disease is the eighteenth cause of deaths worldwide. Despite relatively stable incidences, the prevalence of End-stage renal disease on renal replacement therapy has doubled from 1990 to 2010, and the toll is expected to rise further in the coming decade raising global health concerns. These findings are in line with the reported increase in the global burden of diabetes mellitus and hypertension, the two diseases accounting for the majority of etiologies for End-stage renal disease. The number of diabetes patients worldwide is projected to be 300 million by the year 2025, from 135 million reported in 1995. By 170%, this increase is projected to be more in the developing world as compared to a 42% expected increase in the developed world. Approximately a billion people every year are diagnosed with hypertension, and nearly 7.1 million dies from its complications, including cerebrovascular disease, ischemic heart disease, and End-stage renal disease.

   1.2 Renal replacement therapy:

   Regardless of etiology, patients with ESRD would need renal replacement therapy (RRT) such as hemodialysis, peritoneal dialysis, or a kidney transplant. Hemodialysis and peritoneal dialysis account for initial modalities of renal replacement therapies before renal transplantation is opted. It is predicted that a decade from now, the number of patients on Renal Replacement Therapy (RRT) to be 5439 million worldwide. Of three modalities, renal transplantation is reported to be superior in terms of patients' survival and quality of life. Despite kidney transplant's superiority, hemodialysis is a widely utilized of three renal replacement therapy modalities. It is estimated that of all patients who received RRT in 2008, eighty-nine percent (89%) received hemodialysis. Despite the decrease in the population of ESRD on peritoneal dialysis in developed countries, the number had doubled in ten years by the year 2008 in developing countries.

   1.3 Patients' survival on renal replacement therapy:

   Despite revolutionizing End-stage renal disease treatment, complications associated with renal replacement therapy, and patients' quality of lives worth consideration. Cardiovascular diseases and infections account for significant causes of deaths directly related to dialyzes, while immunosuppression and comorbidities are accounting for substantial causes of fatalities in ESRD patients undergone renal transplant. Other factors predicting mortality include demographic factors, comorbidities, ESRD etiology, nutritional status, and biochemical indices. Caucasians and patients below 45 years have better survival outcomes. Ongoing evidence of inflammation, increased cardiac enzymes, extreme potassium levels, low hemoglobin levels, inadequate dialysis, and lower BMI are associated with poor survival outcomes.

   1.4 RRT challenges in developing countries:

   Access to renal replacement therapies is by far different in developing from the developed world. About 80% of ESRD patients receiving renal replacement therapy worldwide are in developed countries only, meaning it covers only about 12% of the world's population. Though not impossible, the provision of renal replacement therapy in developing countries is challenging. The challenges can range from patient factors like high costs and poor health-seeking behavior, the low budget allocated in non-communicable diseases to technological complexity out of reach of developing countries. Challenges are categorized into three levels of factors, i.e., patient factors; Healthcare and policy and policy factors, and renal registries.

   1.4.1 Patient' factors:

   Adding to the limited coverage of health insurance services, financially constrained patients who constitute a large population of people in developing countries to find it overwhelming to afford high costs of RRT. Furthermore, poor health-seeking behaviors, patients' remoteness, traditional and religious beliefs hinder RRT provision. Literatures report, about 30% of adults are unaware of having hypertension, more than 40% of people with hypertension have not initiated treatment, while 70% of hypertensive patients have not had their hypertension controlled. Also, in some countries, renal transplantation is less often because kidney donation is considered against religious or traditional beliefs.

   1.4.2 Healthcare system factors:

   In most developing countries, renal replacement therapies are centralized in that they are provided at tertiary referral hospitals, which are few for the population they serve, unlike in developed world where satellite hospitals reduce patients load in tertiary hospitals. In Tanzania, for instance, unevenly distributed three public and nine private dialysis offering hospitals serving over fifty-five million residents. In central Tanzania, the first renal replacement facility, UDOM hemodialysis unit was established in 2013, the first renal transplant was done in 2018, collaborating with BMH, and only one kidney transplants have been done ever since. Furthermore, developing countries are still struggling to vaccinate, controlling the spread, and managing past and newly emerging infectious diseases. Increasing incidences and prevalence of non-communicable diseases like ESRD further cripple and deem healthcare budget inadequate.

   1.4.3 Renal registries:

   Only a few African countries have established and organized renal registries. The majority of countries have not had or have failed to maintain them due to several reasons, including financial constraints. This hinders auditing of treatment and quality of care delivery, as well as limiting sources of information and data for researches. This has led developing countries to depend on information and data obtained from developed countries to make significant health decisions. International comparisons of data on ESRD patients and renal replacement therapy may not be correct in terms of validity due to differences in acceptance of the treatment, patients' demographics, socioeconomic burdens, and national health care policies.

   1.5 Research Problem:

   Incidences and prevalence of ESRD have increased in developing countries including, Sub-Saharan African countries. Of different RRT modalities utilized, hemodialysis accounts for the majority. Unlike in developed countries, inadequate renal health facilities, equipment and personnel, insufficient health budget allocation, lack of renal registries, and few published literature regarding hemodialysis in developing countries hinder the provision of hemodialysis to ESRD patients. Furthermore, patient's factors like hemodialysis-treatment costs, poor health-seeking behavior, traditional beliefs, and residency remoteness, further cripple renal replacement therapy provision. Taking Tanzania into account, no renal registry is currently available in the country, leave alone not having any published literature in the region to report short and long-term survival analysis for ESRD patients on maintenance hemodialysis.
2. Methodology

2.1 Data collection and procedure: Patients' information regarding demographics, medical history, physical examination, causes of ESRD, laboratory findings, imaging results, dialysis adequacy, and follow-up will be sought from electronic and physical patients' files. Other information not captured by patients' hospital-record files will be collected separately by the researcher using a separately-designed form. All data will be recorded in a Microsoft Excel spreadsheet and stored in a registry-office computer as well as a backup in OneDrive cloud storage.

2.2 Data Variables:

This study will have dependent and independent variables. The main dependent variable will be death status, classified as nominal (i.e., dead or alive). Other dependent variables were infection (i.e. nominal), hospitalization (i.e. nominal) and time-to-event (i.e. continuous).

Independent variables consisted of both nominal and continuous. These were Age, Sex, ethnicity, smoking status, marital status, education level, health insurance type, residence, comorbidities, employment status, amount of income, duration of illness before referral, initial pulse rate, initial blood pressure, BMI, waist-hip circumference ratio and definitive diagnosis. Other were initial values of Hemoglobin level, total white blood count, platelets level, thyroid-stimulating hormone, serum thyroxine, serum triiodothyronine, serum electrolytes (i.e., potassium, sodium, chloride, magnesium, inorganic phosphates, CO2-combining power, and anion gap), random blood glucose, Liver function tests (Alanine aminotransferases, Aspartate aminotransferases, Total serum protein, serum albumin, total bilirubin, and direct bilirubin and Alkaline phosphatase), muscle enzymes (myoglobin, lactate dehydrogenase, and creatine kinase), urinalysis (albuminuria, proteinuria, urine-pH, glucosuria, urine sedimentation, and 24-hours urine protein). Moreover, initial results for inflammation indices (procalcitonin, erythrocyte sedimentation rate, C-reactive protein, and hypersensitive C-reactive protein), coagulation indices (prothrombin activity, prothrombin time, international normalized ratio, activated partial prothrombin time, thrombin time and d-dimer), lipid profile (low-density lipoprotein, high-density lipoprotein, lipoprotein-alpha, triglycerides, and total cholesterol). Finally, chronic kidney disease stage, type of dialysis catheter, and dialysis adequacy will further be recorded.

2.3 Bias Management:

Bias in this study will be addressed in two levels; study level and outcome level. A potential source of bias foreseen is regarding the patient's record system. UDOM hemodialysis unit utilizes both electronic (newly established) and physical-paper files, meaning every patient will have two records. To eliminate typing errors during feeding data into the electronic system, a registry-officer will extract data from physical-paper files followed by crosschecking with the electronic database by a second registry-officer, for completeness.

To improve data collection accuracy and efficiency, the two dedicated registry-officers will receive one-month training before the official opening of participants' enrollment.

To minimize reporting biases, STROBE checklist-tool (Strengthening the Reporting of Observational Studies in Epidemiology) customized for cohort and case-control studies, will be used in the report write-up of this study.

To minimize publication biases, this protocol is anticipated to be registered to https://clinicaltrials.gov/, before enrollment of participants.

3.4 Data analysis:

Statistical analysis will be done according to the objectives in question. Firstly, predictors of deaths will be identified by binary logistic regression, using death status as a dependent variable and demographics, medical history, clinical picture, and dialysis adequacy as independent variables. Comparisons will be made by odds ratio between predictors and results tested for statistical significance, at 95% using independent t-test. Computer software SPSS will be used. Independent variables showing significant statistical significance to be predicting deaths will be utilized to construct survival curves by Kaplan-Meier. Survival at 1, 3, and 5 years will be deducted from Kaplan-Meier curves and reported. Computer software SAS will be used here.

A descriptive analysis will be conducted to depict common causes of infection and re-hospitalization, their incidences, and prevalence. Time-to-event analysis for first infection and rehospitalization will be constructed using Kaplan-Maier survival curves. Time-to-event comparison between common causes of diseases and rehospitalization will be compared using the log-rank test. All statistical analyses will be done by computer software SPSS, using a 95% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with end-stage renal disease due to any etiology.
* Participants initiated on maintenance dialysis.
* Participants attending Benjamin Mkapa Hospital or UDOM health center.
* Eligible participants consented to participate in the study.

Exclusion Criteria:

* Patients diagnosed with acute kidney injury.
* Patients with CKD stage other than stage 5.
* Patients underwent kidney transplantation.
* Patients on dialysis other than hemodialysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: End stage renal disease patients requiring maintanance hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 5 Years
  To identify predictors for mortality among End-stage renal disease patients undergoing maintenance hemodialysis at UDOM (University of Dodoma) health center and Benjamin Mkapa Hospital using by binary logistic regression.
Survival | 5 Years
  To analyze survival of End-stage renal disease undergoing maintenance hemodialysis at 1, 3 and 5 years, at UDOM health center and Benjamin Mkapa Hospital, using Kaplan-Meier survival curves.

SECONDARY OUTCOMES:
Infection incidence | 5 Years
  To analyze incidences for common causes of infection among End-stage renal disease undergoing maintenance hemodialysis at UDOM health center and Benjamin Mkapa Hospital.
Infection prevalence | 5 Years
  To analyze prevalence of common causes of infection among End-stage renal disease undergoing maintenance hemodialysis at UDOM health center and Benjamin Mkapa Hospital.
Time-to-infection survival | 5 Years
  To analyze time-to-infection survival of common causes of infection among End-stage renal disease undergoing maintenance hemodialysis at UDOM health center and Benjamin Mkapa Hospital, by Kaplan-Maier survival curves.
Incidences of rehospitalization | 5 Years
  To analyze incidences of common causes of rehospitalization among End-stage renal disease undergoing maintenance hemodialysis at UDOM health center and Benjamin Mkapa Hospital.
Prevalence of rehospitalization causes | 5 Years
  To analyze prevalence of common causes of rehospitalization among End-stage renal disease undergoing maintenance hemodialysis at UDOM health center and Benjamin Mkapa Hospital.
Time-to-rehospitalization survival | 5 years
  To analyze time-to-rehospitalization survival in End-stage renal disease patients undergoing maintenance hemodialysis at UDOM health center and Benjamin Mkapa Hospital, by Kaplan-Maier survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Swai, MMed, Principal Investigator — Benjamin Mkapa Hospital
Locations (1):
- Benjamin Mkapa Hospital, Dodoma, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castro A, Neri M, Karopadi AN, Lorenzin A, Marchionna N, Ronco C. How can we advance in renal replacement therapy techniques? Nefrologia (Engl Ed). 2019 Jul-Aug;39(4):372-378. doi: 10.1016/j.nefro.2018.08.012. Epub 2019 Mar 4. English, Spanish. PMID 30846291
- [Background] Obrador GT, Rubilar X, Agazzi E, Estefan J. The Challenge of Providing Renal Replacement Therapy in Developing Countries: The Latin American Perspective. Am J Kidney Dis. 2016 Mar;67(3):499-506. doi: 10.1053/j.ajkd.2015.08.033. Epub 2015 Dec 19. PMID 26709109
- [Background] Almaguer M, Herrera R, Alfonso J, Magrans C, Manalich R, Martinez A. Primary health care strategies for the prevention of end-stage renal disease in Cuba. Kidney Int Suppl. 2005 Aug;(97):S4-10. doi: 10.1111/j.1523-1755.2005.09701.x. PMID 16014098
- [Background] Schena FP. Epidemiology of end-stage renal disease: International comparisons of renal replacement therapy. Kidney International. 2000;57:S39-S45.
- [Background] National High Blood Pressure Education Program. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Bethesda (MD): National Heart, Lung, and Blood Institute (US); 2004 Aug. Report No.: 04-5230. Available from http://www.ncbi.nlm.nih.gov/books/NBK9630/ PMID 20821851
- [Background] Duong CM, Olszyna DP, Nguyen PD, McLaws ML. Challenges of hemodialysis in Vietnam: experience from the first standardized district dialysis unit in Ho Chi Minh City. BMC Nephrol. 2015 Aug 1;16:122. doi: 10.1186/s12882-015-0117-2. PMID 26231882
- [Background] Bello BT, Raji YR, Sanusi I, Braimoh RW, Amira OC, Mabayoje OM. Challenges of providing maintenance hemodialysis in a resource poor country: Experience from a single teaching hospital in Lagos, Southwest Nigeria. Hemodial Int. 2013 Jul;17(3):427-33. doi: 10.1111/hdi.12024. Epub 2013 Feb 3. PMID 23374329
- [Background] Prakash J, Ghosh B, Singh S, Soni A, Rathore SS. Causes of death in renal transplant recipients with functioning allograft. Indian J Nephrol. 2012 Jul;22(4):264-8. doi: 10.4103/0971-4065.101245. PMID 23162269
- [Background] Kansal SK, Morfin JA, Weinhandl ED. Survival and Kidney Transplant Incidence on Home versus In-Center Hemodialysis, Following Peritoneal Dialysis Technique Failure. Perit Dial Int. 2019 Jan-Feb;39(1):25-34. doi: 10.3747/pdi.2017.00207. Epub 2018 Jul 31. PMID 30065065
- [Background] Pauly RP. Survival comparison between intensive hemodialysis and transplantation in the context of the existing literature surrounding nocturnal and short-daily hemodialysis. Nephrol Dial Transplant. 2013 Jan;28(1):44-7. doi: 10.1093/ndt/gfs419. PMID 23300280
- [Background] Wong B, Ravani P, Oliver MJ, Holroyd-Leduc J, Venturato L, Garg AX, Quinn RR. Comparison of Patient Survival Between Hemodialysis and Peritoneal Dialysis Among Patients Eligible for Both Modalities. Am J Kidney Dis. 2018 Mar;71(3):344-351. doi: 10.1053/j.ajkd.2017.08.028. Epub 2017 Nov 22. PMID 29174322
- [Background] Aviles-Gomez R, Luquin-Arellano VH, Garcia-Garcia G, Ibarra-Hernandez M, Briseno-Renteria G. Is renal replacement therapy for all possible in developing countries? Ethn Dis. 2006 Spring;16(2 Suppl 2):S2-70-2. PMID 16774015
- [Background] Li PK, Chow KM. The cost barrier to peritoneal dialysis in the developing world--an Asian perspective. Perit Dial Int. 2001;21 Suppl 3:S307-13. PMID 11887842
- [Background] Mushi L, Marschall P, Flessa S. The cost of dialysis in low and middle-income countries: a systematic review. BMC Health Serv Res. 2015 Nov 12;15:506. doi: 10.1186/s12913-015-1166-8. PMID 26563300
- [Background] Sadler JH. Health promotion for end-stage renal disease patients. Adv Ren Replace Ther. 1998 Oct;5(4):275-85. doi: 10.1016/s1073-4449(98)70019-6. PMID 9792082
- [Background] Meremo AJ, Ngilangwa DP, Mwashambwa MY, Masalu MB, Kapinga J, Tagalile R, Sabi I. Challenges and outcomes of haemodialysis among patients presenting with kidney diseases in Dodoma, Tanzania. BMC Nephrol. 2017 Jul 4;18(1):212. doi: 10.1186/s12882-017-0634-2. PMID 28676037
- [Background] Gupta I, Guin P. Communicable diseases in the South-East Asia Region of the World Health Organization: towards a more effective response. Bull World Health Organ. 2010 Mar;88(3):199-205. doi: 10.2471/BLT.09.065540. PMID 20428387
- [Background] Nyaaba GN, Stronks K, de-Graft Aikins A, Kengne AP, Agyemang C. Tracing Africa's progress towards implementing the Non-Communicable Diseases Global action plan 2013-2020: a synthesis of WHO country profile reports. BMC Public Health. 2017 Apr 5;17(1):297. doi: 10.1186/s12889-017-4199-6. PMID 28381252
- [Background] Davids MR, Caskey FJ, Young T, Balbir Singh GK. Strengthening Renal Registries and ESRD Research in Africa. Semin Nephrol. 2017 May;37(3):211-223. doi: 10.1016/j.semnephrol.2017.02.002. PMID 28532551
- [Background] Jha V, Chugh K. Dialysis in developing countries: Priorities and obstacles2007. 65-71 p.